CLINICAL TRIAL: NCT06280183
Title: The Investigation of the Effects of Functional Inspiratory Muscle Training in Obese Individuals
Brief Title: Functional Inspiratory Muscle Training in Obese Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc.Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 323132
Record Dates: First submitted 2024-01-26; First posted 2024-02-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: obesity; respiratory muscle training; exercise; prevention
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind study three arm study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessor will be blind to the group allocation, and participants will be blind to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic and Resistive Exercise Training (Active Comparator): The exercise program will start with a 5-10 minute warm-up and end with a 5-10 minute cool down. Aerobic exercise is planned at 60-85% of Maximum Heart Rate on the bike for 30-40 minutes.
  Resistive exercise program, covering all major major muscle groups; The upper body (pectoralis, latissimus dorsi, rotator cuff muscles, deltoid, biceps, triceps), abdominal muscles and lower extremities (quadriceps, hamstring, gastrosoleus) will be exercised to strengthen. For upper body muscles, abdominal muscles and lower extremity muscles, 1-3 sets of 10-15 repetitions will be planned as 40-70% of 1 maximum repetition (1RM).
  Interventions: Other: Aerobic+Resistive Exercise Traning
- Functional Inspiratory Muscle Training Group in obese individuals: (Experimental): Inspiratory muscle training will be applied simultaneously with aerobic exercise. This program will create the functional IMT. The exercise program will start with a 5-10 minute warm-up and cool down. Aerobic exercise is planned at 60-85% of MHR on the bike for 30-40 minutes, progress will be achieved. Participants will first work with bicycle ergometry and then continue with IMT in the same session for the first three weeks. The intensity of IMT exercise will be set at 40-60% of MIP. After 10 consecutive breathing cycles, participants will be asked to perform 3-4 breath checks. Resistive exercise program, covering all major muscle groups; The upper body (pectoralis, latissimus dorsi, rotator cuff muscles, deltoid, biceps, triceps), abdominal muscles and lower extremities (quadriceps, hamstring, gastrosoleus) will be exercised to strengthen. For upper body muscles, abdominal muscles and lower extremity muscles, 1-3 sets of 10-15 repetitions will be planned as 40-70% of 1RM.
  Interventions: Other: Functional Inspiratory Muscle Training
- Control Group: (No Intervention): Patient education will be given and no intervention will be made.

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training — Inspiratory muscle training is a technique that combines aerobic training with inspiratory muscle training. will be applied simultaneously with aerobic exercise. Participants will work with bicycle ergometry and then continue with IMT in the same session for the first three weeks. The intensity of IMT exercise will be set at 40-60% of MIP.
  Arms: Functional Inspiratory Muscle Training Group in obese individuals:
Other: Aerobic+Resistive Exercise Traning — Aerobic exercise is planned at 60-85% of the Maximum Heart Rate on a cycle ergometer for 30-40 minutes. Resistive exercise will cover all major muscle groups. The upper body (pectoralis, latissimus dorsi, rotator cuff muscles, deltoid, biceps, triceps), abdominal muscles, and lower extremities (quadriceps, hamstring, gastrosoleus) will be exercised to strengthen. For upper body, abdominal, and lower extremity muscles, 1-3 sets of 10-15 repetitions will be planned as 40-70% of 1 maximum repetition (1RM).
  Arms: Aerobic and Resistive Exercise Training

SUMMARY:
In obese individuals, increased adipose tissue and systemic inflammation play a key role in the development of cardiometabolic diseases, pulmonary system dysfunction, and many respiratory diseases. Existing research has demonstrated beneficial clinical outcomes of inspiratory muscle training or combined aerobic and resistance exercise training in obese individuals. However, this focused on the isolated effects of exercise on obesity. In the current literature, no study is evaluating the effectiveness of functional inspiratory muscle training in obese individuals.

This study aims to investigate the effects of functional inspiratory muscle training on body composition, cardiometabolic markers, functional capacity, respiratory function, respiratory muscle strength, and respiratory muscle performance in obese individuals.

DETAILED DESCRIPTION:
Obesity is characterized by increased adipose tissue and systemic inflammation that play a key role in the development of non-communicable chronic diseases. It is well known that individuals with obesity have decreased exercise capacity and muscle weakness in both peripheral and respiratory muscles.

Exercise training is recommended in addition to healthy dietary habits in managing obesity. Current literature demonstrated beneficial clinical outcomes of isolated inspiratory muscle training or combined aerobic and resistance exercise training in obese individuals.

Functional inspiratory muscle training is a method that combines both aerobic exercise and inspiratory muscle training. In the current literature, no study is evaluating the effectiveness of functional inspiratory muscle training in obese individuals. The aim of this study is to investigate the effect of functional inspiratory muscle training on body composition, cardiometabolic markers, functional capacity, respiratory function, respiratory muscle strength and respiratory muscle performance in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 25-60
* According to the World Health Organization (WHO) classification, those with a body mass index between 30-40 kg/m2
* Volunteering to participate in the research

Exclusion Criteria:

* According to the World Health Organization (WHO) classification, body mass index is over 40 kg/m2
* Functional class III or IV according to the New York Heart Association (NYHA) classification
* Those with a Charlson comorbidity score of 3 and above
* Uncontrolled hypertension, diabetes and unstable angina pectoris
* Cooperative disorders, orthopedic and neurological problems that may interfere with evaluation and treatment
* Individuals with a history of lower extremity-related injury or surgery in the last six months
* Being diagnosed with diabetes and having complications such as nephropathy, retinopathy and neuropathy
* Those with accompanying chronic respiratory disease
* Those with acute infection
* Individuals with middle ear-related pathologies (such as tympanic membrane rupture, otitis)
* Those with a STOP-Bang score of 3 and above
* Individuals with a history of spontaneous or trauma-related pneumothorax
* Smokers
* Pregnancy

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | 10 weeks
  Respiratory muscle strength; It will be evaluated with an intraoral pressure measuring device in a sitting position.
Incremental load test (Respiratory Muscle Endurance) | 10 weeks
  Respiratory muscle endurance will be evaluated by incremental load test. The incremental load test will be performed using the electronic inspiratory loading device (PowerBreathe®-KHP2).
Forced expiratory volume 1st second (Respiratory Function) | 10 weeks
  Spirometric assessment will be performed to determine participants' forced expiratory volume in one second (FEV1).
Forced vital capacity (Respiratory Function) | 10 weeks.
  Spirometric assessment will be performed to determine participants' forced vital capacity (FVC).

SECONDARY OUTCOMES:
Comorbidity Assessment | Day 1
  "Charlson Comorbidity Index" (CMI) will be used to determine the comorbidity levels of obese individuals. The index, which consists of nineteen comorbid diagnosis groups, is a valid method for evaluating chronic diseases and measuring their relationship with mortality. All CMI scores are scored between 0-37. According to the results, 3 levels of comorbidity are defined: low (0), medium (1-2) and high (3+).
Physical Activity Assessment | 10 weeks
  Step Count Measurement: Daily step count will be monitored to determine the physical activity level of the participants. Step count will be assessed with a wearable activity monitor, a portable, easy-to-use tool that can measure objectively (Huawei Watch Fit Special Edition). With its six-axis sensor, the device records the user's physical activity style information in its temporary memory throughout the duration of use. Participants will be asked to wear the activity monitor on their left wrist throughout and only remove it during bathing. After one week of use, the data recorded with the wearable activity monitor will be taken.
Edmonton Obesity Staging System (EOSS) | Day 1
  The Edmonton Obesity Staging System (EOSS) is a five-stage obesity classification system used to determine prognosis and guide treatment when assessing obesity-related risk.
Functional Capacity | 10 weeks
  Submaximal functional exercise capacity of the participants will be evaluated with the six-minute walk test.
Peripheral Muscle Strength | 10 weeks
  M. Quadriceps muscle strength and hand grip strength measurement will be used to evaluate peripheral muscle strength. Hand-held dynamometer will be used to evaluate quadriceps muscle strength and hand grip strength.
Waist circumference | 10 weeks
  Waist circumference will be measured at belly level with the patient in an upright position during expiration, with both feet bearing equal weight.
Hip circumference | 10 weeks
  Hip circumference will be measured at the level of the greater femoral trochanter, with the patient in an upright position, with both feet bearing equal weight.
Body fat-muscle ratios | 10 weeks
  These measurements will be determined by bioelectrical impedance.
Glucose profile | 10 weeks
  Glucose profile after 12 hours of fasting will be measured
Lipid profile | 10 weeks
  Lipid profile after 12 hours of fasting will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akinci, Assoc. Prof., Study Chair — Biruni University; Alihan Oral, Assoc. Prof., Study Director — Biruni University Hospital; Safak Yigit, MSc, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No